CLINICAL TRIAL: NCT06209775
Title: Impact of Perioperative Body Composition Abnormalities on Patient Outcomes After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Shulan (Hangzhou) Hospital (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2023-ZJU-OBS5
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Liver Transplantation; Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Split liver transplantation group: Between January 1, 2015 and December 31, 2022, all recipients who underwent split liver transplantation at the First Affiliated Hospital of the Zhejiang University School of Medicine, Shulan (Hangzhou) Hospital and the Affiliated Hospital of Qingdao University were considered for inclusion. After exluding pediatric cases, multiorgan transplantations, liver cancer patients with macrovascular invasion or distant metastasis and recipients without computed tomography (CT) scan within three months before split liver transplantation, 240 patients were included. The procedures of organ donation and transplantation were strictly implemented under the regulation of the China Organ Donation Committee (CODC), Organ Transplant Committee (OTC) and the Declaration of Helsinki (as revised in 2013). All donor livers came from donation after citizens' death and there was no procurement from prisoners.
- Whole liver transplantation group: 2991 patients received deceased donor liver transplantation (DDLT) for liver cancers in the First Affiliated Hospital of Zhejiang University School of Medicine (Hangzhou, China) between January 2015 and January 2021, Shulan (Hangzhou) Hospital (Hangzhou, China) between July 2017 and January 2021, and the Affiliated Hospital of Qingdao University between January 2015 and January 2022. The subject selection process is shown in Figure 1. After excluding transplants for benign disease (N=1667), pediatric transplants (N=141), re-transplants (N=219), multi-organ transplants (N=23), transplants for neoplasms other than HCC (N=62), patients with macrovascular invasion (N=159), patients who died within 30 days after transplantation (N=55), patients with incomplete clinical data (N=45), and patients without pre-LT CT scans (N=208), 756 patients were studied.

SUMMARY:
Accumulating evidence suggests the prognostic significance of body composition in chronic diseases and neoplastic diseases. CT imaging-based body composition abnormalities are significantly associated with post-LT adverse outcomes including decreased quality of life (QOL), impaired graft regeneration and mortality. However, the perioperative changes in body composition and their potential clinical implications remain unexplored. The objective of this study is to systematically explore and clarify the correlation between body composition and the prognosis of liver transplant patients through dynamic peri-transplant mornitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing deceased donor liver transplantation (DDLT) for the first time.

Exclusion Criteria:

* Pediatric transplants
* Re-transplants
* Multi-organ transplants
* Liver cancer patients with macrovascular invasion or distant metastasis
* Patients who died within 30 days after transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liver transplant patients from 3 transplant centers in China
Sampling Method: Non-Probability Sample
Enrollment: 996 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative mortality | 2015.1.1-2022.12.31
Postoperative recurrence of liver cancer | 2015.1.1-2022.12.31

REFERENCES:
- [Derived] Chen H, Hu Z, Xu Q, He C, Yang X, Shen W, Lin Z, Li H, Zhuang L, Cai J, Lerut J, Zheng S, Lu D, Xu X. The adverse impact of perioperative body composition abnormalities on outcomes after split liver transplantation: a multicenter retrospective cohort study. Int J Surg. 2024 Jun 1;110(6):3543-3553. doi: 10.1097/JS9.0000000000001303. PMID 38489552